CLINICAL TRIAL: NCT02194569
Title: Magnesium Balance of Citrate-based Continuous Venovenous Hemofiltration, Effect of Citrate Dose.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Willem Boer, MD, Ziekenhuis Oost-Limburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CIDOUT
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Critically Ill; Acute Kidney Injury
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury | interventions — Citric Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High citrate group (Experimental): Blood flow according to weight.Target citrate concentration is 4,5 mmol/L blood flow delivered as prismocitrate 18/0 pre-filter. After correction for filtration fraction, the required further amount of substitution fluid is given post filter to achieve a hemofiltration rate of 30 ml/kg/hr. Blood citrate concentrations are tailored to achieve an iCa of 0.8-1.1 mg/dL.
  Interventions: Drug: Citrate
- Low citrate group (Experimental): Blood flow according to weight. Target citrate concentration is 2.5 mmol/L blood flow delivered as prismocitrate 18/0 pre-filter. After correction for filtration fraction, the required further amount of substitution fluid is given post filter to achieve a hemofiltration rate of 30 ml/kg/hr. Blood citrate concentrations are tailored to achieve an iCa of 1.3-1.6 mg/dL.
  Interventions: Drug: Citrate

INTERVENTIONS:
Drug: Citrate

SUMMARY:
Rationale:

A higher citrate dose during continuous venovenous hemofiltration provides better anticoagulation but possibly a higher risk of citrate accumulation in case of metabolic limitations. A higher citrate dose also increases magnesium loss in ultrafiltrate, while a negative magnesium balance is unwanted.

Objective:

Aim of this study is to determine the magnesium balance of citrate-based continuous veno-venous hemofiltration (CVVH) and to determine whether and to which extent the magnesium balance depends on citrate dose.

Study design and methods:

A prospective randomized study conducted in critically ill patients with acute kidney injury (AKI), treated with CVVH, with either low dose citrate (2.5 mmol/L blood flow in the filter) or high dose citrate (4.5 mmol/L blood flow in the filter) as anti-coagulant, targeting a postfilter ionized Calcium (iCa) of resp. 1.3-1.6 mg/dL (0.325-0.4 mmol/L) and 0.8-1.1 mg/dL (0.2-0.275 mmol/L). Post-filter blood as well as effluent aliquots and bloodconcentrations in the patient are tested for the following variables:

(0 , 2 , 4, 6, 12 and 24 hrs): Total Magnesium (tMg) and total Calcium (tCa), ionized Ca (iCa)(bloodgas analyzer). In addition, hematocrit, albumin, total protein, ureum and creatinine and parathormone (PTH) are determined in arterial blood at 0 and 24 hrs or at the time of protocol exit and citrate concentrations in postfilter and arterial blood at 1 and 24 hrs or at protocol exit.

Sample sites: arterial line, postfilter port (after postdilution and calcium compensation), effluent sample. All flow rates to be noted.

Study population:

Twenty patients admitted to intensive care, requiring continuous renal replacement therapy (CRRT) for AKI.

Intervention:

Anti-coagulation with either low dose citraat (2.5 mmol/L blood flow) or high dose citraat (4.5 mmol/L blood flow) targeting postfilter iCa of resp. 1.3-1.6 and 0.8-1.1 mg/dL. Both regimens are within standard protocolled CVVH treatment in the intensive care department.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients requiring CRRT for AKI (RIFLE criteria)
* Written informed consent from the patient or legal representative

Exclusion Criteria:

* pre-existing chronic renal insufficiency requiring dialysis
* chronic immunosuppression
* liver cirrhosis Child-Pugh C
* severe or shock-related hepatitis
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-07; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Mg balance of CVVH treatment | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Willem Boer, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost Limburg, Genk, Limburg, Belgium

REFERENCES:
- [Derived] Boer W, Fivez T, Vander Laenen M, Bruckers L, Gron HJ, Schetz M, Oudemans-van Straaten H. Citrate dose for continuous hemofiltration: effect on calcium and magnesium balance, parathormone and vitamin D status, a randomized controlled trial. BMC Nephrol. 2021 Dec 11;22(1):409. doi: 10.1186/s12882-021-02598-2. PMID 34895160
- [Derived] Tsujimoto H, Tsujimoto Y, Nakata Y, Fujii T, Takahashi S, Akazawa M, Kataoka Y. Pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2020 Dec 14;12(12):CD012467. doi: 10.1002/14651858.CD012467.pub3. PMID 33314078